CLINICAL TRIAL: NCT03801421
Title: Mass Continuous Suture With PDS Versus Interrupted Suture With Thread on Major Abdominal Incision: A Randomized Controlled Trial
Brief Title: Mass Continous Suture With PDS Versus Interrupted Suture With Thread on Major Abdominal Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Zhang Xu-Feng, Professor, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AFCRC2017SJ-007-2
Record Dates: First submitted 2019-01-06; First posted 2019-01-11 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Surgical Wound; Suture, Complication
Keywords: Surgical Wound; Suture, Complication
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continous suture group (Experimental): The surgical incision will be treated by mass continous suture with PDS.
  Interventions: Procedure: Mass continous suture with PDS
- Control group (Active Comparator): The surgical incision will be treated by interrupted suture with thread.
  Interventions: Procedure: Interrupted suture with thread

INTERVENTIONS:
Procedure: Mass continous suture with PDS — The surgical incision will be treated by mass continous suture with PDS.
  Arms: Continous suture group
Procedure: Interrupted suture with thread — The surgical incision will be treated by interrupted suture with thread.
  Arms: Control group

SUMMARY:
A better suture technology will reduce postoperative incision complications. This study is designed to compare mass continous suture with PDS and interrupted suture with thread on major abdominal incision.

DETAILED DESCRIPTION:
A better suture technology will reduce postoperative incision complications. The previous retrospective cohort study from the investigator has demonstrated that continuous mass suture with PDS led to shorter incision closure time, early wound healing and comparable incisional complications versus interrupted thread suture. As such, the current RCT study will include 100 subjects with major abdominal incision. They will be divided into two groups randomly: Mass suture gorup, mass continuous suture with PDS, Control group, interrupted suture with thread. The wound healing time, stitches removal time and incidence of incision complications will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* the patient with major abdominal incision.
* the incision is longer than 10 cm
* aged between 18 to 65 years old

Exclusion Criteria:

* Pregnant woman
* Patient with diabetes
* Patient with a history of cardiovascular disease, including coronary heart disease and stroke.
* Severe lung diseases such as COPD and asthma
* Patients undergoing emergent or infectious surgery
* Patients with surgical site infection
* No autonomy, inability or unwillingness to participate in follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
healing time, d (day) | Up to 1 month after surgery
  Time duration between the date of surgery to the date of stitches off

SECONDARY OUTCOMES:
incidence of incision complications | Up to 1 month after surgery
  The incision complications include infection, dehiscence, fat liquefaction, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Xu-Feng Zhang, MD, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China